CLINICAL TRIAL: NCT03712358
Title: A Phase I Trial of PVSRIPO for Patients With Unresectable Melanoma
Brief Title: PVSRIPO for Patients With Unresectable Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed to enrollment due to business decision prior to enrolling Cohort 4
Sponsor: Istari Oncology, Inc. (Industry)
Collaborators: Duke University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00090774; K08CA237726 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 0 (PVSRIPO) (Experimental): A single dose of PVSRIPO into a single lesion.
  Interventions: Biological: PVSRIPO
- Cohort 1 (PVSRIPO) (Experimental): A single dose of PVSRIPO into 2 different lesions, 21 days apart, when applicable per dose escalation guidelines.
  Interventions: Biological: PVSRIPO
- Cohort 2 (PVSRIPO) (Experimental): A single dose of PVSRIPO into 3 different lesions, 21 days apart, when applicable per dose escalation guidelines.
  Interventions: Biological: PVSRIPO
- Cohort 3 (PVSRIPO) (Experimental): A single dose of PVSRIPO into 3 different lesions, 21 days apart, when applicable per dose escalation guidelines.
  Interventions: Biological: PVSRIPO
- Cohort 4 (PVSRIPO) (Experimental): A single dose of PVSRIPO into a single lesion, followed by PVSRIPO injected into up to 6 lesions at Day 10 and every 21 days thereafter.
  Interventions: Biological: PVSRIPO

INTERVENTIONS:
Biological: PVSRIPO — Intralesional injection of PVSRIPO.

SUMMARY:
This study is a Phase I study of oncolytic polio/rhinovirus recombinant (PVSRIPO) to primarily characterize the safety and tolerability of PVSRIPO in patients with AJCC Stage IIIB, IIIC, or IV melanoma in a modified 3+3 phase 1 trial design. Lesion biopsies and blood samples will be obtained pre- and post-injection throughout the study for routine histology/molecular genetic testing and immunologic analysis, respectively. Exploratory objectives include describing the response rates of PVSRIPO-injected versus non-injected lesion(s), the number of CD8 positive T cells present in the tumor biopsies before and after injection of PVSRIPO, and after PVSRIPO administration: the pathologic response in tumor biopsies, changes in the tumor microenvironment, and how systemic immune cell populations may change.

DETAILED DESCRIPTION:
The Primary Objective of the study is to determine the safety profile of PVSRIPO in Stage IIIB, IIIC, and IV recurrent melanoma patients as determined by dose-limiting toxicities (DLT) by cohort, as well as in those retreated with PVSRIPO, when PVSRIPO is injected intralesionally into 1 to 3 or more cutaneous or subcutaneous lesions. As planned, up to 18 patients may be treated with PVSRIPO.

Biopsy material will be obtained from tumor tissue prior to and following virus administration, which may be subjected to routine histology along with molecular genetic testing and evaluation of pathological response. Whole blood for immunologic analyses will also be collected throughout the study period.

Routine study visits will occur through Day 126. Thereafter, visits will occur every 2-3 months for up to 2 years for subjects who do not progress. For patients with progressive disease, chart review only will occur every 3 months starting at the time of progression.

Patients who previously participated in Cohorts 0 through 3, who in the opinion of the investigator, may benefit from continued PVSRIPO administration, may be eligible to receive additional injections.

ELIGIBILITY:
Inclusion Criteria:

1. Undergone prior vaccination against PV and received a boost immunization with trivalent IPOL® (Sanofi-Pasteur SA) at least 1 week, but less than 6 weeks, prior to administration of PVSRIPO (within 6 months of PVSRIPO retreatment).

   a. Note: Patients who are unsure of their prior vaccination status/who have not been vaccinated must provide proof of vaccination and/or evidence of anti-PV immunity prior to enrollment, as applicable.
2. The patient must have received a boost immunization with trivalent inactivated IPOL™ (Sanofi-Pasteur) at least 1 week prior to administration of the study agent.
3. Patient must have histologically proven unresectable, recurrent, melanoma, stage IIIB, IIIC, or stage IV (AJCC staging must be documented in patient's medical record, as determined by CT of the chest, abdomen and pelvis, and/or whole body positron emission tomography (PET) scan, and MRI of the brain within 4 weeks prior to administration of study drug).
4. Patients with BRAF mutations, must have failed at least 2 lines of therapy, specifically one BRAF targeted therapy and at least one anti-PD-1 based therapy. For BRAF wild type, patients must have failed at least one anti-PD-1 based therapy.
5. Patient must be ≥ 18 years of age.
6. Patient must have an Eastern Cooperative Oncology Group (ECOG) / Zubrod status of 0-1.
7. Patient's disease must be bi-dimensionally measurable by caliper or radiological method as defined in the immune-related response criteria (irRC).
8. At least 1 injectable cutaneous, subcutaneous or nodal melanoma lesion ≥ 10 mm in longest diameter or, multiple injectable melanoma lesions which in aggregate have a longest diameter of ≥ 10 mm (Cohorts 0 and possibly 1). For cohorts where 2 or 3 injections are planned (Cohorts 1 and 2), the patient must have at least 2 injectable melanoma lesions (when 2 doses are planned) or ≥3 injectable melanoma lesions when at least 3 doses are planned in different lesions (Cohorts 2 through 4).

   a. Note: PVSRIPO retreatment requires ≥2 lesions amenable to injection.
9. At least one measurable lesion that will not be injected.
10. Serum lactate dehydrogenase (LDH) levels less than 1.5 x upper limit of normal (ULN).
11. Patient must have adequate bone marrow, liver and renal function as assessed by the following:

    1. Hemoglobin > 9.0 g/dl
    2. White blood count (WBC) of > 2000 m3
    3. Absolute neutrophil count (ANC) > 1,000/mm3
    4. Platelet count > 75,000/mm3
    5. Total bilirubin < 2.0 x ULN
    6. Alanine aminotransferse (ALT) and aspartate aminotransferance (AST) < 2.5 x the ULN

Exclusion Criteria:

1. Females who are pregnant or breast-feeding.
2. Adults of reproductive potential not employing an effective method of birth control.
3. Patients with severe, active co-morbidity, defined as follows:

   1. Patients with an active infection requiring treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C).
   2. Patients with impaired cardiac function or clinically significant cardiac disease, such as congestive heart failure requiring treatment (New York Heart Association Class ≥ 2), uncontrolled hypertension or clinically significant arrhythmia; QTcF > 470 msec on ECG if performed or congenital long QT syndrome; acute myocardial infarction or unstable angina pectoris < 3 months prior to study.
   3. Patients with known lung (FEV1 < 50%) disease or uncontrolled diabetes mellitus (HgbA1c>7).
   4. Patients with albumin allergy.
   5. Autoimmune disease: History of or current active autoimmune diseases, [e.g. including but not limited to inflammatory bowel diseases [IBD], rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (such as Guillain-Barre syndrome)]. Vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are not exclusionary.
   6. Known immunosuppressive disease, human immunodeficiency virus (HIV) infection, or chronic Hepatitis B or C.
4. Patients with a previous history of neurological complications due to PV infection.
5. Patients who have not recovered from the toxic effects of prior chemo- and/or radiation therapy. Guidelines for this recovery period are dependent upon the specific therapeutic agent being used. Toxicities must have resolved to CTCAE grade 1 or less with the following exceptions (alopecia, fatigue, vitiligo).
6. Patients with undetectable anti-tetanus toxoid IgG.
7. Patients with known history of agammaglobulinemia.
8. Patients on greater than 10 mg per day of prednisone within the 2 weeks prior to admission for PVSRIPO injection.
9. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups).
10. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin.
11. Clinically active cerebral or bone metastases.
12. Greater than 3 visceral metastases (this does not include nodal metastases associated with visceral organs).
13. Prior allogeneic stem cell transplantation.
14. Concomitant therapy with any of the following: IL-2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses). However, during the course of the study, use of corticosteroids is allowed if used for treating immune related adverse events (irAE), adrenal insufficiencies, or if administered at doses of prednisone 10 mg daily or equivalent.
15. Active clinically serious infection > CTCAE Grade 2.
16. Antineoplastic therapy, radiotherapy, or any other investigational drug within 15 days prior to first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Franklin, Study Director — Istari Oncology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Brown MC, Beasley GM, McKay ZP, Yang Y, Desjardins A, Randazzo DM, Landi D, Ashley DM, Bigner DD, Nair SK, Gromeier M. Intratumor childhood vaccine-specific CD4+ T-cell recall coordinates antitumor CD8+ T cells and eosinophils. J Immunother Cancer. 2023 Apr;11(4):e006463. doi: 10.1136/jitc-2022-006463. PMID 37072349
- [Derived] Beasley GM, Brown MC, Farrow NE, Landa K, Al-Rohil RN, Selim MA, Therien AD, Jung SH, Gao J, Boczkowski D, Holl EK, Salama AKS, Bigner DD, Gromeier M, Nair SK. Multimodality analysis confers a prognostic benefit of a T-cell infiltrated tumor microenvironment and peripheral immune status in patients with melanoma. J Immunother Cancer. 2022 Sep;10(9):e005052. doi: 10.1136/jitc-2022-005052. PMID 36175036
- [Derived] Beasley GM, Nair SK, Farrow NE, Landa K, Selim MA, Wiggs CA, Jung SH, Bigner DD, True Kelly A, Gromeier M, Salama AK. Phase I trial of intratumoral PVSRIPO in patients with unresectable, treatment-refractory melanoma. J Immunother Cancer. 2021 Apr;9(4):e002203. doi: 10.1136/jitc-2020-002203. PMID 33875611

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 0 (PVSRIPO): A single dose of 1.0 x 10^8 TCID50 PVSRIPO into a single lesion.
  PVSRIPO: Intralesional injection of PVSRIPO.
- Cohort 1 (PVSRIPO): A single dose of 1.0 x 10^8 TCID50 PVSRIPO into 2 different lesions, 21 days apart, when applicable per dose escalation guidelines.Total dose 2.0 x 10^8 TCID50.
  PVSRIPO: Intralesional injection of PVSRIPO.
- Cohort 2 (PVSRIPO): A single dose of 1.0 x 10^8 TCID50 PVSRIPO into 3 different lesions, 21 days apart, when applicable per dose escalation guidelines. Total dose 3.0 x 10^8 TCID50.
  PVSRIPO: Intralesional injection of PVSRIPO.
- Cohort 3 (PVSRIPO): A single dose of 1.0 x 10^8 TCID50 PVSRIPO into 3 different lesions, 21 days apart, when applicable per dose escalation guidelines. Total dose of 3.0 x 10^8 TCID50 PVSRIPO.
  PVSRIPO: Intralesional injection of PVSRIPO.
- Cohort 4 (PVSRIPO): A single dose of 1.0 x 10^8 TCID50 PVSRIPO into a single lesion, followed by PVSRIPO injected into up to 6 lesions at Day 10 and every 21 days thereafter.
  PVSRIPO: Intralesional injection of PVSRIPO.
Period: Overall Study
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Started | 3 | 3 | 3 | 3 | 0
Completed | 3 | 3 | 3 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study closed to enrollment due to business decision prior to enrolling Cohort 4.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (10.69) | 59.7 (19.55) | 70.3 (4.62) | 71.0 (7.81) |  | 65.4 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 |  | 4
  Male | 2 | 1 | 3 | 2 |  | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 |  | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 |  | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 | 0 |  | 0
  White | 3 | 3 | 3 | 3 |  | 12
  More than one race | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Dose Limiting Toxicity by Cohort
Description: To characterize the safety and tolerability of PVSRIPO in American Joint Committee on Cancer (AJCC) Stage IIIB, IIIC, or IV melanoma.
Time Frame: 24 months
Population: Study closed to enrollment due to business decision prior to enrolling Cohort 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0
Participants | 0 | 0 | 0 | 0 |

2. Other Pre Specified Outcome: Response Rates Via Measurement of Cutaneous Lesions Every 3 Weeks
Description: To describe the response rates via lesion size of PVSRIPO-injected versus non-injected lesion(s) as defined per the investigator using immune related response criteria (irRC).
Time Frame: 24 months
Population: Based on immune-related response criteria (irRC).
Measure: Number; unit: participants
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0
participants
  Not Evaluable | 3 | 3 | 1 | 1 |
  immune-related Partial Response (irPR) | 0 | 0 | 2 | 1 |
  immune related Stable Disease (irSD) | 0 | 0 | 0 | 1 |

3. Other Pre Specified Outcome: Number of CD8 Positive T Cells by Immunohistochemistry on Pre Treatment and Post Treatment Biopsy (Cohorts 0-3 Only)
Description: To describe the number of CD8 positive T cells present in the tumor biopsies before and after injection of PVSRIPO.
Time Frame: 4.1 months
Population: Cohort 4 not enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0
Participants
  Pre-treatment: Absent | 0 | 0 | 0 | 0 | 0
  Pre-treatment: Sparse | 3 | 0 | 0 | 0 | 0
  Pre-treatment: Dense | 0 | 3 | 1 | 0 | 0
  Pre-treatment: Missing data | 0 | 0 | 2 | 3 | 0
  Post-treatment: Absent | 0 | 0 | 0 | 0 | 0
  Post-treatment: Sparse | 2 | 1 | 1 | 0 | 0
  Post-treatment: Dense | 0 | 2 | 1 | 0 | 0
  Post-treatment: Missing data | 1 | 0 | 1 | 3 | 0

4. Other Pre Specified Outcome: The Change in Tumor Pathology From Baseline to After PVSRIPO Injection
Description: Determine the pathologic response in tumor biopsies after PVSRIPO by confirming presence or absence of viable tumor cells.
Time Frame: 4.1 months
Population: Insufficient sample for analysis and Cohort 4 not enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 0
Participants
  No response | 2 | 2 | 1 | 0 | 0
  Complete response | 0 | 0 | 1 | 1 | 0
  Missing data | 1 | 1 | 1 | 2 | 0

5. Other Pre Specified Outcome: The Detection of Viral Replication in Injected Versus Non Injected Lesions (Cohorts 0-3 Only)
Description: Determine viral replication via a number of methods (e.g., qRT-PCR, ICH).
Time Frame: 4.1 months
Population: Insufficient sample for analysis and Cohort 4 not enrolled
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: The Change in Inflammatory Cells and Markers After PVSRIPO in Injected Versus Non Injected Lesions (Cohorts 0-3 Only)
Description: Determine changes in the tumor microenvironment from biopsies after PVSRIPO; includes but not limited to examination of CD8, PVR (CD155), PD-L1, CD4, FoxPE, and PD-1.
Time Frame: 4.1 months
Population: Data were not collected for this measure
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Change Relative to Baseline in Type and/or Function of T Cells Via Flow Cytometry (Cohorts 0-3 Only)
Description: Describe how systemic immune cell populations may change after treatment with PVSRIPO.
Time Frame: 24 months
Population: Cohort 3 missing data; Cohort 4 not enrolled
Measure: Mean (Full Range); unit: cells per 200,000 events
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
cells per 200,000 events
  Pre-treatment | 10315 [799 to 18923] | 7879 [725 to 13932] | 39776 [10557 to 86395] |  |
  Post-treatment | 5949 [903 to 10996] | 20574 [9452 to 31697] | 102332 [55708 to 148957] |  |

ADVERSE EVENTS:
Time Frame: From signing the informed consent form until the participant's end of study visit, up to 2 years
Description: The # of participants at risk in Cohort 4 is zero because the study closed to enrollment due to business decision prior to enrolling Cohort 4.
Arm/Group | Cohort 0 (PVSRIPO) | Cohort 1 (PVSRIPO) | Cohort 2 (PVSRIPO) | Cohort 3 (PVSRIPO) | Cohort 4 (PVSRIPO)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 0 (PVSRIPO) (N=3) | Cohort 1 (PVSRIPO) (N=3) | Cohort 2 (PVSRIPO) (N=3) | Cohort 3 (PVSRIPO) (N=3) | Cohort 4 (PVSRIPO) (N=0)
pruritis (General disorders) | 1 | 2 | 2 | 2 | 0
erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 1 | 0
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
incisional drainage (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
rash macro-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03712358/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03712358/SAP_001.pdf